CLINICAL TRIAL: NCT04940507
Title: Safety and Feasibility of Focused Ultrasound-enabled Liquid Biopsy in Patients With Brain Tumours
Brief Title: BRAINFUL (BRAIN Tumor Focused Ultrasound-enabled Liquid Biopsy) Trial
Acronym: BRAINFUL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Brain Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20-6243; 707126 (Other Grant/Funding Number: Canadian Cancer Society and Brain Canada Foundation)
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Brain Neoplasms; Liquid Biopsy
Keywords: High-Intensity Focused Ultrasound Ablation
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tumor cohort (Experimental): Intervention 1:
  Participants will undergo a partial tumor ablation with MRgFUS using ExAblate Neuro 4000 device (InSightec Ltd, Tirat Carmel, Israel). Blood and CSF samples will be drawn on several timepoints before and after the procedure.
  Intervention 2:
  Participants will undergo a standard of care tumor biopsy/excision one day after the "Intervention 1". Blood samples will be drawn on several timepoints before and after the procedure.
  Interventions: Procedure: Magnetic Resonance Guided Focused Ultrasound Tumor Ablation and Liquid Biopsy Acquisition
- Essential tremor cohort (Other): To identify the levels of circulating free DNA release after MRgFUS procedure in non-tumoral patients and to check whether the MRgFUS procedure induce tumoral mutations itself, we will draw blood samples from essential tremor patients before and after standard of care MRgFUS thalamotomy procedure.
  Interventions: Procedure: Magnetic Resonance Guided Focused Ultrasound Thalamotomy

INTERVENTIONS:
Procedure: Magnetic Resonance Guided Focused Ultrasound Tumor Ablation and Liquid Biopsy Acquisition — Partial ablation of tumor using ExAblate Neuro 4000 device (InSightec Ltd, Tirat Carmel, Israel) and blood and CSF draws for liquid biopsy
  Other Names: Neurosurgical Tumor Biopsy/Excision
  Arms: Tumor cohort
Procedure: Magnetic Resonance Guided Focused Ultrasound Thalamotomy — Ablation of VIM nucleus of thalamus with MRgFUS using ExAblate Neuro 4000 Device (InSightec Ltd, Tirat Carmel, Israel) and blood draws.
  Arms: Essential tremor cohort

SUMMARY:
Background:

Accessing brain tumor material for pathological diagnosis requires invasive procedures that carry risk to patients including brain hemorrhages and death. Liquid biopsies are emerging non-invasive alternatives to direct tumour biopsies but the abundance of circulating tumor DNA (ctDNA) is relatively low and this limits our ability to accurately make the molecular diagnosis of brain tumors. We have recently shown promising results that suggest that the analysis of blood samples can distinguish brain tumor types. We now want to couple liquid biopsies with high intensity focused ultrasound (HIFU) to enhance the release of tumor DNA into the circulation and increase the sensitivity/and specificity of liquid biopsies for brain tumors. The aim of this project is to build on our preliminary findings and investigate the the time dependent changes associated with HIFU of a tumor to see if it improves accuracy of diagnosis and specifically molecular subtyping of tumors based on peripheral blood and cerebrospinal fluid (CSF) circulating tumor derived markers following HIFU.

DETAILED DESCRIPTION:
Objective:

To increase plasma ctDNA and thereby improve the identification of ctDNA-based genomic and epigenomic biomarkers, magnetic resonance-guided focused ultrasound (MRgFUS) will be utilized in brain tumor patients to enhance the release of tumour DNA into blood circulation and CSF.

Study type:

Single-center, prospective, single-blinded, single arm, controlled clinical trial.

Experimental Approach:

Aim 1: To assess the utility of MRgFUS in enhancing the abundance of brain tumor ctDNA. Non-invasive brain tumor diagnosis and treatment has the potential to transform patient care but necessitates improved sensitivity for epigenomic and genomic biomarker detection than is possible with current approaches. It has been shown that MRgFUS can enhance circulating biomarker presence in animal models and that it can be safely utilized intracranially in humans. Accordingly, this Aim expands on existing literature to utilize MRgFUS to improve the abundance of circulating tumour DNA in brain tumor patients as the first step in the transformation to non-invasive diagnosis and monitoring. The results of this aim will inform on the optimal timepoint of plasma sampling after MRgFUS to obtain the highest quantity of ctDNA for use in molecular analyses.

Aim 2: To evaluate the utility of MRgFUS in enhancing the non-invasive detection of brain tumor methylation signatures. Published work from our lab has shown that gliomas can be distinguished from other brain tumours accurately using the sensitive detection of plasma methylation alterations (mean AUC 0.99). Unfortunately, the identification of glioma subtype is more limited, and the models developed to distinguish glioblastomas have a mean AUC of 0.71 (only for IDH). Given that glioblastomas have a distinct biology and are typically managed differently than lower grade gliomas, the ability to non-invasively determine glioma subtype is clinically very important. The use of MRgFUS to improve the sensitivity of non-invasive plasma methylation signature detection of brain tumors in this aim has the potential to change care for these patients by allowing for either avoidance of surgery in patients who are not amenable to resection, improved surgical planning for those that are, and longitudinal repeat sampling to identify clonal evolution and acquisition of new clinically-relevant molecular alterations.

Aim 3: To improve the non-invasive detection of brain tumor genomic alterations using MRgFUS. Attempts to identify tumour genomic alterations non-invasively through blood samples has largely been ineffective due to the low ctDNA abundance and its short half-life. The identification of tumoral mutations is important for prognostication at the time of diagnosis and to identify alterations with available targeted treatments. This aim utilizes MRgFUS to improve ctDNA abundance in order to allow for non-invasive detection of clinically-relevant genomic alterations such as IDH1/2, TERT promoter, CDKN2A/B, PTEN, EGFR, TP53, BRAF, and PDGFRA mutations in glioblastoma patients.

Significance:

Overall, this work will support the use of a MRgFUS-enhanced liquid biopsy approach that avoids the risks of intracranial biopsy and identifies genomic and epigenomic alterations of brain tumors with higher sensitives and specificities than can be achieved with current plasma-based approaches which approach the accuracy of tissue-based approaches. This non-invasive identification of brain tumor methylation signatures will allow for diagnosis without the need for invasive intracranial biopsy. Additionally, non-invasive identification of and monitoring for genomic alterations in brain tumors will be important for treatment decision, particularly for targeted treatments typically offered at the time of recurrence which depend on mutations found in the tumor.

The overarching goal of this project is to shift the paradigm of ascertaining brain tumor diagnosis from high-risk invasive procedures to a non-invasive diagnostic approach with potentially additional advantages, such as reaching surgically inaccessible brain regions, capturing the tumoral heterogeneity, serial monitoring of the tumor, early detection of progressive disease and distinguishing tumor from pseudoprogression/radiation necrosis.

Impact Statement Liquid biopsies in brain tumor patients are limited to date by low or even undetectable levels of tumor biomarkers. We hypothesize that this limitation can be overcome by a novel approach using high intensity focused ultrasound to significantly increase the release tumor biomarker into the blood and thereby improve the sensitivity of liquid biopsy. This work is expected to lead to a paradigm shift in the way we approach brain tumour diagnosis and treatment, allowing for non-invasive patient prognostication and treatment target identification to optimize approach to prevent glioblastoma progression. We expect many changes to neuro-oncology care to follow as approaches to improve liquid biopsy improve as outlined below.

Firstly, a common indication for surgery in brain tumour patients is for a tumour biopsy, as treatment decisions for other cancer therapies like radiotherapy and systemic therapies depend on tumour diagnosis and specific tumour mutations which cannot be made based on imaging alone. For these patients, it is expected that non-invasive diagnosis would replace the need for neurosurgical biopsy and avoid associated risks including hemorrhage and death. Additionally, for patients who require surgery for tumour removal together with diagnosis, the ability to diagnose tumour prior to surgery will inform preoperative and intraoperative decision making regarding the aggressiveness of tumour resection undertaken.

Additionally, the median time to glioblastoma recurrence is 7-8 months and treatment decision making at the time of recurrence typically leads to the use of targeted treatments, often in the context of clinical trials, which requires repeat tumour biopsies. Not only will this technology avoid the need for repeat biopsies at the time of recurrence in these patients and associated risks, but this technology also allows for the entirety of tumoral heterogeneity to be assessed for genomic/epigenomic alterations and not only the small portion of tumour biopsied neurosurgically which may not be representative to the overall tumour heterogeneity.

Not only does this approach avoid the need for tumour re-biopsy at the time of recurrence, but it would allow for ongoing longitudinal tumour sampling during routine clinical follow-up which is not possible with neurosurgical biopsies but is possible using non-invasive technology alone as is done here. This can be used to model tumour response to treatment, allowing for early identification of resistance mechanisms, while also tracking clonal evolution over time and outside of when surgical biopsies are indicated. Longitudinal MRgFUS-enhanced liquid biopsy is also expected to allow for the early diagnosis of tumor progression by distinguishing it from pseudoprogression/radiation necrosis, which is an important differential diagnosis.

In addition to the diagnostic benefits, spatially partial thermocoagulation necrosis of the tumor after MRgFUS procedure may contribute to the treatment of the patients by cytoreduction of the viable tumor cells and a decrease in their invasion capacity. This is particularly of concern to patients with surgically unresectable tumors in eloquent areas and will benefit these patients significantly. It is also expected that MRgFUS-induced hyperthermia in tumours may enhance the efficacy of radiation treatment. We may potentially simultaneously radiosensitize tumor while obtaining liquid biopsies to monitor treatment response and track of clonal evolution over time.

In summary, this study is unique in pairing experts with both MRgFUS experience and non-invasive liquid tumour biopsy expertise, in order to apply the benefits of MRgFUS to a new clinical problem that has the potential to change the way we diagnose and monitor glioblastoma patients. Currently, patients require invasive neurosurgical procedures to diagnose glioblastoma that have associated risks and complications. Our lab has shown that liquid biopsy techniques can be utilized in brain tumour diagnostics but low abundance of circulating tumour DNA limits our ability to determine tumour subtypes and mutations non-invasively. The enhancement of circulating tumour DNA after MRgFUS is a unique approach to improving the sensitivity and specificity of non-invasive approaches to identify glioblastoma epigenomic and genomic alterations. The results of this work may lead change in the way we manage glioblastoma patients, moving away from invasive diagnostic procedures and towards non-invasive tumour diagnosis and monitoring to guide treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* New MRI-diagnosed intracranial lesions that are suitable to biopsy surgically
* The lesion to be treated is clearly defined and can be well distinguished from surrounding brain tissue.
* Male or female aged 18 years or older
* Capable of providing informed consent and complying with study procedures, including tolerability in the supine position and MRI examination without significant claustrophobia, and acceptance of surgery (open or stereotactic) after HIFU treatment.
* Able to communicate during the ExAblate® MRgFUS procedure.
* Karnofsky rating 70-100

Exclusion Criteria:

* If region of treatment locates in < 1.0 cm from the inner table of the skull, on skull base or in the posterior fossa
* Presence of hydrocephalus, severe vomiting, intractable headache or decreased level of consciousness due to increased intracranial pressure
* Unable to complete high-density CT and MRI studies of the head at the any other MRI contraindication, such as:

  * Large body habitus and not fitting comfortably into the scanner
  * Difficulty lying supine and still for up to 2 in the MRI unit or significant claustrophobia
* MRI findings:

  * Active infection/inflammation
  * Acute or chronic brain haemorrhages
  * Moderate/severe brain edema or midline shift >15 mm
* Clips or other metallic implanted objects in the skull or the brain, except shunts
* Significant cardiac disease or unstable hemodynamic status.
* On medications that increase the bleeding risk, specifically: a) aspirin or another antiplatelet medication (clopidogrel, prasugrel, ticlopidine, abciximab) for the last 7 days prior to treatment; b) oral, subcutaneous or intravenous anticoagulant medications, such as oral vitamin K inhibitors for the last 7 days, non-vitamin K inhibitor oral anticoagulant (dabigatran, apixaban, rivaroxaban) for the last 72 hours, and intravenous or subcutaneous heparin-derived compounds for the last 48 hours
* Abnormal coagulation profile, specifically: platelet <100,000/μl, Prothrombin Time >14 seconds, activated partial thromboplastin time (aPTT) >36 seconds, and INR > 1.3
* Unqualified fit for the anaesthesia by an anesthesiologist assessment, ASA IV-V.
* Currently in a clinical trial involving an investigational product or non-approved use of a drug or device.
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood and CSF levels of the circulating free DNA | Pre-MRgFUS: Within 1 hour; Post-MRgFUS: Within 1 hour, between 3-4 hours; Pre-surgery: Within 1 hour; Post-surgery:Within 1 hour, between 16-24 hours
  Difference in concentration of cfDNA between the blood and CSF samples acquired before and after MRgFUS

SECONDARY OUTCOMES:
The optimal time-point of liquid biopsy acquisition | Pre-MRgFUS: Within 1 hour; Post-MRgFUS: Within 1 hour, between 3-4 hours; Pre-surgery: Within 1 hour; Post-surgery:Within 1 hour, between 16-24 hours
  by understanding the time of highest plasma cfDNA concentration by the comparison of the cfDNA concentrations across all time-points after the MRgFUS procedure
Safety (procedure-related complications) | Post-MRgFUS: Within 1 hour, between 3-4 hours; Pre-surgery: Within 1 hour; Post-surgery: Within 1 hour, between 16-24 hours and 1 month
  incidence of adverse events as assessed by clinical examination during surgery and at 1-month follow-up
Epigenomic analysis | Pre-MRgFUS: Within 1 hour; Post-MRgFUS: Within 1 hour, between 3-4 hours; Pre-surgery: Within 1 hour; Post-surgery:Within 1 hour, between 16-24 hours
  Involves detection of DNA methylation signatures of tumours and application of set of models to discriminate them. Impact of MRgFUS will assessed by the change in AUC values of brain tumor classification models in MRgFUS treated patients, comparing plasma and CSF samples obtained prior to and after the procedure
Genomic analysis | Pre-MRgFUS: Within 1 hour; Post-MRgFUS: Within 1 hour, between 3-4 hours; Pre-surgery: Within 1 hour; Post-surgery:Within 1 hour, between 16-24 hours
  Involves detection of relevant tumoral gene mutations. For tumour group, we will compute the concordance of plasma and CSF based genomic alteration targeted sequencing results with tissue-based results. For control group, we will compare the baseline and post-procedure tumoral gene mutations to understand FUS cause de novo tumoral mutations.

CONTACTS AND LOCATIONS:
Overall Officials: Andres M. Lozano, MD, PhD, Principal Investigator — University of Toronto; Gelareh Zadeh, MD, PhD, Principal Investigator — University of Toronto
Locations (1):
- Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No